CLINICAL TRIAL: NCT02847039
Title: Early Repolarization Syndrome: Define the Risk, Stratify the Coverage and Understand the Causes - Clinical and Genetic Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/09/62
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Early Repolarization Syndrome
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Early repolarization syndrome: Patients with an aspect of early repolarization syndrome or belonging to a family in which the diagnosis of early repolarization was identified.
  Interventions: Genetic: Blood samples

INTERVENTIONS:
Genetic: Blood samples — Blood samples at baseline.

SUMMARY:
The research project aims to try to answer the many questions raised by the identification of new early repolarization syndrome. The questions are varied with both taking optimal clinical management of patients, the frequency and significance of this anomaly in the population on the electrophysiological and molecular basis responsible for this electrocardiographic abnormality.

To try to answer these many questions, the approach will be twofold: clinical and genetic.

* Establishment of a clinical database containing information of patients who have been identified as carriers of the anomaly based on the initial clinical presentation in order to determine their prognoses.
* Physiological approach will be based on a molecular approach to identify genetic abnormalities may be involved in this syndrome.
* 200 asymptomatic patients and an unlimited number of patients who presented syncope or aborted sudden death will be included.

A blood sample (15 ml) will be performed at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Presence of early repolarization aspect, determined by the J point elevation of at least 0.1 mV above the isoelectric line, with or without extra-ST segment elevation in at least two leads and / or lateral.
* Parameters ECG D2 level of the bypass measurable for the presence of long QT syndrome.
* Late potentials ventricular analyzable.
* For patients with ventricular fibrillation, negative search for other causes of ventricular fibrillation.
* For patients with syncope, clinical assessment should included at a minimum, performing a cardiac ultrasound and a stress test.

Exclusion Criteria:

* Impossibility to receive clear information (patient's intellectual default).
* Refusal to sign the informed consent for participation.
* Under protective measure of justice.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with an aspect of early repolarization syndrome or belonging to a family in which the diagnosis of early repolarization was identified.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ventricular fibrillation or sudden death | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France